CLINICAL TRIAL: NCT01141972
Title: The Role of Vitamin D in Menopause: Relationship to Menopausal Symptoms in Body Composition
Acronym: FLASH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Pro00001445
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Hot Flushes; Menopause, Premature; Obesity; Vitamin D Deficiency
Keywords: Vitamin D; Obesity; Menopause; Hot Flashes
MeSH Terms: conditions — Hot Flashes; Menopause, Premature; Obesity; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplement (Active Comparator): We will administer 100,000 IU Vitamin D3 orally as an observed 1-time bolus and then prescribe 1000 IU by mouth daily. These doses have achieved sufficiency in other populations.99, 100 We will use the level of sufficiency (≥30 ng/ml [≥75 nmol/L]) that is recommended by most experts in the field.89-91, 93, 95, 96, 101-105 We will repeat the bolus at 1 month if the target level is not achieved. The control group will receive matching placebo and a similar proportion will go through a dummy titration. All women consuming less than 800 mg/day of calcium (by dietary history) will receive 500 mg of calcium to ensure sufficiency
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Current standard of practice does not dictate that otherwise healthy early menopausal women have Vitamin D levels evaluated. Women with Vitamin D levels between 10 and 29 ng/ml who receive placebo will be receiving usual care (i.e., no additional Vitamin D repletion above intake at the time of screening).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — We will administer 100,000 IU Vitamin D3 orally as an observed 1-time bolus and then prescribe 1000 IU by mouth daily. These doses have achieved sufficiency in other populations.99, 100 We will use the level of sufficiency (≥30 ng/ml [≥75 nmol/L]) that is recommended by most experts in the field.89-91, 93, 95, 96, 101-105 We will repeat the bolus at 1 month if the target level is not achieved. The control group will receive matching placebo and a similar proportion will go through a dummy titration. All women consuming less than 800 mg/day of calcium (by dietary history) will receive 500 mg of calcium to ensure sufficiency.
  Arms: Supplement
Other: Placebo — Current standard of practice does not dictate that otherwise healthy early menopausal women have Vitamin D levels evaluated. Women with Vitamin D levels between 10 and 29 ng/ml who receive placebo will be receiving usual care (i.e., no additional Vitamin D repletion above intake at the time of screening).
  Arms: Placebo

SUMMARY:
Specific Aim 1: To compare effects of Vitamin D supplementation to usual care on symptoms in women transitioning to early postmenopause and determine the associated effect size in order to conduct a power analysis for a future RCT. Hypothesis: Vitamin D insufficient women in early postmenopause who are randomized to supplementation, titrated to achieve sufficiency for 2 months, will have fewer symptoms including hot flashes, mood, and musculoskeletal complaints than women randomized to usual care.

Specific Aim 2: To compare effects of Vitamin D supplementation to usual care on body composition (by dual-energy x-ray absorptiometry [DXA] and by weight, BMI, waist to hip ratio) in overweight/obese women transitioning to early postmenopause and determine the associated effect size for a power analysis for a future RCT. Hypothesis: Vitamin D insufficient women in the menopausal transition randomized to supplementation, titrated to achieve sufficiency for 9 months, will improve DXA body composition (less total body and abdominal fat), compared to women in usual care, who will have increased body weight, including total and abdominal fat.

Specific Aim 3: To estimate the proportion of overweight/obese middle-aged women who achieve sufficiency by 1 month versus 2 or more months and to determine if achieving sufficiency by 1 month varies by baseline characteristics. Hypothesis: About 80% of participants will achieve sufficient Vitamin D level by 1 month. Those who need more than 1 month for sufficiency will have lower baseline levels and higher initial BMI.

DETAILED DESCRIPTION:
It is increasingly recognized that Vitamin D deficiency affects more than just bone health. Links between Vitamin D deficiency have been established or purported for diabetes, the metabolic syndrome, cardiovascular disease, and cancer. We propose to explore if Vitamin D replacement (safe, readily available, and inexpensive) has beneficial effects on 2 novel outcomes in early postmenopausal women: menopause-related symptoms and body composition.

Most women transitioning through menopause, especially those with higher percent body fat, will experience hot flashes through a mean of 4 to 5 years. Many also have mood disturbances and muscle aches although the link with the menopausal transition is less clear. In many, these symptoms are severe enough to negatively impact their quality of life, work performance, and interpersonal relationships. Current treatments for menopause-related symptoms, such as menopausal hormone therapy, antidepressants, and anticonvulsants, have significant side effects and serious long term adverse consequences and symptoms recur after treatment discontinuation. A safe, inexpensive, well-tolerated treatment is therefore of high priority.

Both our preliminary data in early postmenopausal women and a 2010 publication of women on aromatase inhibitors for breast cancer show an association between Vitamin D deficiency and menopause-related symptoms including hot flashes. It is postulated that a contributor to hot flashes is a menopausal decline in serotonin, a neurotransmitter with known effects on thermoregulation. As Vitamin D can protect against experimental serotonin depletion in rats, one proposed mechanism for symptom alleviation is prevention of serotonin decline in menopause.

Both Vitamin D deficiency and the menopausal transition are associated with mood disturbances and musculoskeletal aches. Because estrogen increases the activity of the enzyme responsible for activating Vitamin D, the fall in estrogen that occurs during the menopausal transition could uncover previously subclinical Vitamin D deficiency. Indeed, Vitamin D can improved mood and muscle aches in non-menopausal populations, but its effects in menopausal women, where the benefits may be magnified, have not been previously studied.

ELIGIBILITY:
Inclusion Criteria:

* Women in late menopausal transition or early menopause
* Age 40-55
* BMI >25 kg/m2
* Suffer from menopausal symptoms
* Change in previously regular cycles consisting of at least ≥2 skipped cycles and an interval of amenorrhea (≥60 days) in the last year
* Negative pregnancy test
* Vitamin D insufficiency (<30 ng/ml)
* Weight stability (+/- 5%) for 3 months

Exclusion Criteria:

* No period for >12 months
* Hormone use (i.e. menopausal hormone therapy, oral contraceptive, other hormonal medications) in last 3 months
* History of hysterectomy more than 11 months ago
* Abnormal screening blood tests (i.e. elevated serum calcium level, elevated creatinine)
* History of medical conditions where Vitamin D supplementation is not indicated (i.e. chronic renal insufficiency, elevated calcium, sarcoidosis or other granulomatous disease, lymphoma, or tuberculosis
* History of osteoporosis or osteoporosis on baseline DXA (expect less than 4% of screened population)84
* Vitamin D deficiency (<10 ng/ml) as we felt it was unethical to withhold supplementation for 12 months in severe deficiency (according to our KPNW survey, this will exclude <2% of population)
* Consuming more than 400 IU of Vitamin D supplementation daily (we felt such doses taken outside of the study design could confound results)
* Current smoker (within the last year)
* Taking medications that affect body weight
* Prior bariatric surgery
* Taking medications or herbal supplements that affect mood (i.e. antidepressants) or menopausal symptoms (i.e. herbal meds) or sleep
* Weighing more than 400 pounds (cannot fit on DEXA scan)
* Not fluent in English or cognitively impaired

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
compare effects of Vitamin D supplementation to usual care on symptoms in women transitioning to early postmenopause and determine the associated effects | 12 months
  Vitamin D levels will be measured at baseline, after dose adjustments, and at the 3 month and final visit.

SECONDARY OUTCOMES:
compare effects of Vitamin D supplementation to usual care on body composition (by dual-energy x-ray absorptiometry [DXA] and by weight, BMI, waist to hip ratio) in overweight/obese women transitioning to early postmenopause | 12 months
  Body composition will be measured with DXA113, 114 and anthropometric techniques (weight, height, BMI, waist to hip ratio)

CONTACTS AND LOCATIONS:
Overall Officials: Erin S. LeBlanc, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States